CLINICAL TRIAL: NCT05039593
Title: The Effect of Oral Care Frequency on Oral Mucosa Membrane Integrity in Patients With Mechanical Ventilation Support
Brief Title: Oral Care Frequency in Mechanically Ventilated Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Aslıhan Tahtali Turgut, Nurse, Aydin Adnan Menderes University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: Oral Care Frequency
Record Dates: First submitted 2021-07-02; First posted 2021-09-09 (Actual); Last update posted 2022-07-20 (Actual); Status verified 2022-07

CONDITIONS: Oral Complications
Keywords: Oral care; Chlorhexidine; Mechanical Ventilation
MeSH Terms: interventions — Chlorhexidine

STUDY DESIGN:
Intervention Model Description: Before starting the practice in this study, the purpose of the research will be explained to all nurses working in the unit by the researchers and an information meeting about oral care will be held. After the operability of the guide in the intensive care unit is ensured, the data collection phase will begin. Randomization of patients will be done by the nurse in charge of the service.
  The frequency of oral care of the patients will be in three groups. Oral care will be done twice a day for the patients in the first group, 3 times a day for the patients in the second group, and 4 times a day for the patients in the third group. Oral care of the patients will be applied according to the guide used in the training given to the nurses.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- first group (Experimental): The patients in the first group will be given oral care with 0.12% chlorhexidine twice a day.
  Interventions: Other: chlorhexidine
- second group (Experimental): The patients in the second group will be given oral care with 0.12% chlorhexidine 3 times a day.
  Interventions: Other: chlorhexidine
- third group (Experimental): The patients in the third group will be given oral care with 0.12% chlorhexidine 4 times a day.
  Interventions: Other: chlorhexidine

INTERVENTIONS:
Other: chlorhexidine — The population of the research is the patients hospitalized in the Internal Medicine intensive care unit of Aydın Adnan Menderes University Practice and Research Hospital between 01.06.2021 and 01.06.2022, and the sample is; Patients who are older than 18 years of age, who are in the first 24 hours of mechanical ventilation, who are 18 years of age and older, and whose relatives have consented.Oral care of the patients will be done with 0.12% chlorhexidine solution, and the frequency of oral care will be in three groups. Oral care will be done twice a day for the patients in the first group, 3 times a day for the patients in the second group, and 4 times a day for the patients in the third group. Oral care of the patients will be applied according to the guide used in the training given to the nurses.

SUMMARY:
Many problems may develop in patients due to mechanical ventilation in intensive care units. These include ventilator-associated pneumonia, decreased cerebral perfusion, venous air embolism, sinus and eye infections, neuromuscular dysfunctions and skin sores may be seen in intensive care patients undergoing mechanical ventilation. If adequate oral hygiene is not provided in patients on mechanical ventilation support, dry mouth, halitosis, disruption of tissue integrity in and around the mouth, intraoral infections and periodontal diseases may occur. Most importantly, ventilator-associated pneumonia (VIP) may develop in patients dependent on mechanical ventilation due to deficient oral care.

Chlorhexidine solution is widely used in oral care. However, there is a need for evidence about the frequency of oral care with which chlorhexidine solution on oral mucous membrane integrity in patients under mechanical ventilation support. Oral care frequency was not examined in these existing studies. Therefore, this study was planned to determine the effect of three different oral care frequencies on the integrity of the oral mucous membrane in patients connected to mechanical ventilators.

DETAILED DESCRIPTION:
Oral hygiene is one of the applications where the individual needs the most hygienic care. Providing oral care and maintaining oral hygiene improves the comfort and quality of life by ensuring that the individual eats healthy and feels well.Inadequate oral care can negatively affect all these, as well as cause problems such as dry mouth, dental caries, periodontal diseases, bad breath and stomatitis.Therefore, in order to maintain oral health, individuals must perform oral care effectively.

Nurses need to have adequate oral intake to maintain the integrity of the oral mucosa, especially in patients who cannot be fed orally, with fluid restriction, administered nasogastric tube, mouth breathing, receiving oxygen therapy, undergoing oral and maxillofacial surgery, undergoing radiation therapy, chemotherapy, in the terminal period, in coma, and in patients dependent on mechanical ventilator. care must be provided.

Defense mechanisms in intensive care patients are affected by their disease and multiple interventions that circumvent natural host defenses. Treatments applied in intensive care units, lack of fluid intake of the patient, and some materials used for treatment and care cause changes in the oral mucous membrane. Inadequate protective mechanisms in patients can lead to both local and systemic complications such as caries, periodontal disease, oral mucosal infections, and ventilator-associated pneumonia.

Bacterial oropharyngeal colonization progressively changes to tracheal colonization leading to ventilator-associated pneumonia.

Especially in patients connected to mechanical ventilators, the entry of bacteria into the respiratory tract is facilitated and increased due to the endotracheal tube, causing the coughing reflex and mucociliar activity to be impaired and secretion to increase. In this case, gram-positive bacteria that make up the normal flora in the oral mucosa are replaced by gram-negative bacteria, causing changes in the oral flora and plaque formation on the teeth. Therefore, oral care becomes much more important.The solution and frequency to be used gain importance for oral care to be effective on the integrity of the oral mucous membrane.

In the literature, it is recommended to use chlorhexidine gluconate solution in oral care to prevent the development of ventilator-associated pneumonia in mechanically ventilated patients.However, there is no evidence on how often oral care should be performed.

When the literature is reviewed, further studies with conclusive evidence to show how often chlorhexidine gluconate is effective are needed. For this reason, this study was planned to determine the effect of three different oral care frequencies on the integrity of the oral mucous membrane in patients dependent on mechanical ventilators.

The research is planned to be carried out between 01.06.2021 and 01.06.2022 in the internal medicine intensive care unit of Aydın Adnan Menderes University Practice and Research Hospital.

The population of the research is the patients hospitalized in the Internal Medicine intensive care unit of Aydın Adnan Menderes University Practice and Research Hospital between 01.06.2021 and 01.06.2022, and the sample is; Patients who are older than 18 years of age, who are in the first 24 hours of mechanical ventilation, who are 18 years of age and older, and whose relatives have consented. The sample of the research; Patients with thrombocytopenia, leukopenia and oral aphthae, stomatitis, candiasis, gingivitis who have had an oral surgical procedure will not be accepted.

Before starting the practice in this study, the purpose of the research will be explained to all nurses working in the unit by the researchers and an information meeting about oral care will be held. After the operability of the guide in the intensive care unit is ensured, the data collection phase will begin. Randomization of patients will be done by the nurse in charge of the service.

The frequency of oral care of the patients will be in three groups. Oral care will be done twice a day for the patients in the first group, 3 times a day for the patients in the second group, and 4 times a day for the patients in the third group. Oral care of the patients will be applied according to the guide used in the training given to the nurses. In oral care, 0.12% chlorhexidine solution will be used.

The concentration of 0.12% of the chlorhexidine gluconate solution planned to be used in the research is the most frequently used form compared to the other concentrations of the solution. And no side effects were noted in the studies.

For this reason, 0.12% chlorhexidine solution was preferred. When the literature is examined, this density was preferred because it is the most frequently used solution in the oral care of patients under mechanical ventilation support.

The oral mucosa of the patients will be evaluated with the Oral Evaluation Scale by the researcher before the first oral care application every morning for four days. According to the score obtained from the scale, the researcher will evaluate the patients as normal oral mucosa, mild dysfunction, moderate dysfunction and severe dysfunction.

ELIGIBILITY:
Inclusion Criteria:

* who are over 18 years old,
* In the first 24 hours of mechanical ventilation,
* It will consist of patients with consent from their relatives.

Exclusion Criteria:

* Surgery for the mouth,
* Patients with oral aphthae, stomatitis, candiasis, gingivitis will not be taken.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2021-07-05 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

PRIMARY OUTCOMES:
Oral mucosal evaluation of patients. | Oral care is given to patient groups 2 times a day, 3 times a day, 4 times a day for 4 days. Evaluation will be done at the beginning of the study and every day for 4 days.
  The oral mucosa of the patients will be evaluated with the Eilers Mouth Rating Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Gülengün Türk, Prof.Dr, Study Director — Aydın Adnan Menderes University, Faculty of Nursing, Department of Nursing Fundamentals
Locations (1):
- Aydın Adnan Menderes University, Aydin, Efeler, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] La Combe B, Maherault AC, Messika J, Billard-Pomares T, Branger C, Landraud L, Dreyfuss D, Dib F, Massias L, Ricard JD. Oropharyngeal Bacterial Colonization after Chlorhexidine Mouthwash in Mechanically Ventilated Critically Ill Patients. Anesthesiology. 2018 Dec;129(6):1140-1148. doi: 10.1097/ALN.0000000000002451. PMID 30247201
- [Background] Villar CC, Pannuti CM, Nery DM, Morillo CM, Carmona MJ, Romito GA. Effectiveness of Intraoral Chlorhexidine Protocols in the Prevention of Ventilator-Associated Pneumonia: Meta-Analysis and Systematic Review. Respir Care. 2016 Sep;61(9):1245-59. doi: 10.4187/respcare.04610. Epub 2016 Aug 9. PMID 27507174
- [Background] Deschepper M, Waegeman W, Eeckloo K, Vogelaers D, Blot S. Effects of chlorhexidine gluconate oral care on hospital mortality: a hospital-wide, observational cohort study. Intensive Care Med. 2018 Jul;44(7):1017-1026. doi: 10.1007/s00134-018-5171-3. Epub 2018 May 9. PMID 29744564
- [Background] Kocacal Guler E, Turk G. Oral Chlorhexidine Against Ventilator-Associated Pneumonia and Microbial Colonization in Intensive Care Patients. West J Nurs Res. 2019 Jun;41(6):901-919. doi: 10.1177/0193945918781531. Epub 2018 Jun 15. PMID 29907077
- [Background] Haghighi A, Shafipour V, Bagheri-Nesami M, Gholipour Baradari A, Yazdani Charati J. The impact of oral care on oral health status and prevention of ventilator-associated pneumonia in critically ill patients. Aust Crit Care. 2017 Mar;30(2):69-73. doi: 10.1016/j.aucc.2016.07.002. Epub 2016 Aug 4. PMID 27499527
- [Background] Houston S, Hougland P, Anderson JJ, LaRocco M, Kennedy V, Gentry LO. Effectiveness of 0.12% chlorhexidine gluconate oral rinse in reducing prevalence of nosocomial pneumonia in patients undergoing heart surgery. Am J Crit Care. 2002 Nov;11(6):567-70. PMID 12425407
- [Background] Lee S, Lighvan NL, McCredie V, Pechlivanoglou P, Krahn M, Quinonez C, Azarpazhooh A. Chlorhexidine-Related Mortality Rate in Critically Ill Subjects in Intensive Care Units: A Systematic Review and Meta-Analysis. Respir Care. 2019 Mar;64(3):337-349. doi: 10.4187/respcare.06434. PMID 30850551
- [Background] McCue MK, Palmer GA. Use of Chlorhexidine to Prevent Ventilator-Associated Pneumonia in a Long-term Care Setting: A Retrospective Medical Record Review. J Nurs Care Qual. 2019 Jul/Sep;34(3):263-268. doi: 10.1097/NCQ.0000000000000367. PMID 30325851
- [Background] Ory J, Raybaud E, Chabanne R, Cosserant B, Faure JS, Guerin R, Calvet L, Pereira B, Mourgues C, Guelon D, Traore O. Comparative study of 2 oral care protocols in intensive care units. Am J Infect Control. 2017 Mar 1;45(3):245-250. doi: 10.1016/j.ajic.2016.09.006. Epub 2016 Oct 27. PMID 28341071
- [Background] Saddki N, Mohamad Sani FE, Tin-Oo MM. Oral care for intubated patients: a survey of intensive care unit nurses. Nurs Crit Care. 2017 Mar;22(2):89-98. doi: 10.1111/nicc.12119. Epub 2014 Oct 28. PMID 25349099
- [Background] Turk G, Kocacal Guler E, Eser I, Khorshid L. Oral care practices of intensive care nurses: a descriptive study. Int J Nurs Pract. 2012 Aug;18(4):347-53. doi: 10.1111/j.1440-172X.2012.02045.x. PMID 22845634
- [Background] Zand F, Zahed L, Mansouri P, Dehghanrad F, Bahrani M, Ghorbani M. The effects of oral rinse with 0.2% and 2% chlorhexidine on oropharyngeal colonization and ventilator associated pneumonia in adults' intensive care units. J Crit Care. 2017 Aug;40:318-322. doi: 10.1016/j.jcrc.2017.02.029. Epub 2017 Mar 1. PMID 28320561
- [Result] Bordenave C. [Evaluation of the effectiveness of a protocol of intensification of mouth care (teeth brushing and chlorhexidine 0.12%) on the colonisation of tracheal aspirations in intubated and ventilated patients in intensive care]. Rech Soins Infirm. 2011 Sep;(106):92-8. French. PMID 21972580